CLINICAL TRIAL: NCT02065544
Title: Remission Rates of New Type 2 Diabetes With Weight Loss and Exercise
Acronym: Resolution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Philip Ades, Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS: M11-198
Record Dates: First submitted 2014-02-11; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; behavioral weight loss; exercise training; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- behavioral weight loss and exercise (Experimental): weight loss and exercise lifestyle intervention over a 6 month period
  Interventions: Behavioral: behavioral weight loss and exercise

INTERVENTIONS:
Behavioral: behavioral weight loss and exercise — Weight loss and exercise counseling

SUMMARY:
This is a study of the effects of weight loss and exercise training on glucose control as measured by the Hemoglobin A 1 C in individuals with recently diagnosed Type 2 Diabetes. Study outcomes are measured at 6 months. The primary outcome is the HBA1c at 6-months. Secondary outcomes include body weight, fitness, lipid profiles and HS-CRP, a measure of inflammation. The study hypothesis is that the program of weight loss and exercise will put >50% of individuals into "remission" of their type 2 Diabetes as measured by a HBA1c of < 6.5%.

DETAILED DESCRIPTION:
This is a study of the effects of weight loss and exercise training on glucose control as measured by the Hemoglobin A 1 C in individuals with recently diagnosed Type 2 Diabetes. Study outcomes are measured at 6 months. The primary outcome is the HBA1c at 6-months. Secondary outcomes include body weight, fitness, lipid profiles and HS-CRP, a measure of inflammation. The study hypothesis is that the program of weight loss and exercise will put >50% of individuals into "remission" of their type 2 Diabetes as measured by a HBA1c of < 6.5%.

The study replicates the clinical situation where selected patients with new type 2 diabetes, who are motivated to try an intensive lifestyle intervention, might replicate our study intervention if we are able to show a high remission rate (e.g. > 50%) for individuals in the study.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of type 2 diabetes since 12 months
* BMI>27
* HBA1c > 6.5, , 8.0

Exclusion Criteria:

* HBA1c >8.0
* BMI< 27

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6-months
  HBA1c was the primary outcome as a measure of glucose control in individuals with recently diagnosed type 2 diabetes.

SECONDARY OUTCOMES:
lipid profile | 6 months
  A lipid profile will be drawn before, and after the 6 month intervention
HS-C Reactive Protein | 6 months
  A HS-C Reactive Protein will be drawn before and after the 6 month intervention.
Aerobic Fitness | 6 months
  Aerobic fitness will be measured as Peak Vo2 on the treadmill before and after the 6 month intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Ades, MD, Principal Investigator — University of Vermont